CLINICAL TRIAL: NCT00290511
Title: A Phase II Study of R-FND, Followed by Zevalin Radioimmunotherapy, and Subsequent Maintenance Rituximab for Advanced Stage Follicular Lymphoma With High-Risk Features
Brief Title: Rituximab, Fludarabine, Mitoxantrone, Dexamethasone (R-FND) Plus Zevalin for High-Risk Follicular Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry); Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0287; NCI-2011-02453 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Results first posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-03

CONDITIONS: Lymphoma
Keywords: Follicular Lymphoma; Zevalin; Ibritumomab Tiuxetan; IDEC-Y2B8; Fludarabine; Fludara; Dexamethasone; Mitoxantrone; Rituximab; Rituxan; R-FND; Fludarabine Phosphate; Decadron
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — fludarabine; fludarabine phosphate; Mitoxantrone; Rituximab; ibritumomab tiuxetan; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- R-FIND + Zevalin (Experimental): Fludarabine 25 mg/m^2 intravenous (IV) over 5-30 minutes on Days 2-4. Mitoxantrone 10 mg/m^2 IV over 5-30 minutes on Day 2. Rituximab 375 mg/m^2 IV over 4-6 hours on Day 1 and 8; maintenance Rituximab = 375 mg/m^2 IV over 4-6 hours on Day 1 only, a single dose every other month for 12 months (6 doses total). Zevalin 0.3 mCi/kg IV after 4 cycles of R-FND. Dexamethasone 20 mg by mouth (PO) or IV daily on Days 2-6.
  Interventions: Drug: Fludarabine; Drug: Mitoxantrone; Drug: Rituximab; Drug: Zevalin; Drug: Dexamethasone

INTERVENTIONS:
Drug: Fludarabine — 25 mg/m^2 intravenous (IV) over 5-30 minutes on Days 2-4.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Mitoxantrone — 10 mg/m^2 IV over 5-30 minutes on Day 2.
  Other Names: Novantrone
Drug: Rituximab — 375 mg/m^2 IV over 4-6 hours on Day 1 and 8; maintenance Rituximab = 375 mg/m^2 IV over 4-6 hours on Day 1 only, a single dose every other month for 12 months (6 doses total).
  Other Names: Rituxan
Drug: Zevalin — 0.3 mCi/kg IV after 4 cycles of R-FND.
  Other Names: Ibritumomab Tiuxetan; IDEC-Y2B8
Drug: Dexamethasone — 20 mg by mouth (PO) or IV daily on Days 2-6.
  Other Names: Decadron

SUMMARY:
The goal of this clinical research study is to learn if chemotherapy given with rituximab, followed by Ibritumomab tiuxetan (Zevalin), and then followed by rituximab can help to control lymphoma. The safety of this treatment schedule will also be studied.

Objectives:

1. To assess whether the time to progression for these high-risk patients can be prolonged to a median of 36 months, compared to the historical expectation of approximately 24 months.
2. To assess the tolerance and efficacy of Y2B8 (Zevalin) after R-FND (rituximab, fludarabine, mitoxantrone, dexamethasone) in patients with high-risk stage III-IV follicular lymphoma
3. To assess overall response, failure-free survival, and survival of this strategy compared to our historical experience with FND (fludarabine, mitoxantrone, dexamethasone) alone or R-FND
4. To assess the tolerance and efficacy of maintenance therapy with rituximab.
5. To maximize the 12-month molecular remission rate for patients with high-risk stage III-IV follicular lymphoma
6. to correlate the results of quantitative PCR assay with classical PCR and with clinical outcome

DETAILED DESCRIPTION:
The treatments used in this program include several standard chemotherapy agents (fludarabine, mitoxantrone, and dexamethasone). Also, immune therapy agents will be given, including rituximab (a monoclonal antibody that attacks B-cells, which is what this type of lymphoma is made of), and Ibritumomab tiuxetan (another similar monoclonal antibody, which delivers radiation to the lymphoma cells to strengthen the attack).

You will receive rituximab on Days 1 and 8 of the first cycle, and on Day 1 only of Cycles 2-4 of the monthly cycles of chemotherapy, called R-FND. R-FND includes rituximab and fludarabine, mitoxantrone, and dexamethasone. Fludarabine will be given for 3 days, mitoxantrone for 1 day, and dexamethasone for 5 days of each 28-day cycle (FND). After 4 cycles of R-FND, you will receive Ibritumomab tiuxetan. After the Ibritumomab tiuxetan, you will receive rituximab every 2 months for 1 year. All are given by vein. Sometimes dexamethasone can be given in pill form.

During the study, you will have blood tests (about 2 tablespoons), sometimes every week. Every 2 cycles, you will have a chest x-ray and CT scans of the abdomen and pelvis. Bone marrow samples will be taken. Heart function tests will be done as needed.

If you desire, it may be possible for you to receive some of your study treatment at home (from your home doctor). Your study doctor will discuss this possibility with you. If this is the case, your home doctor will receive a letter telling him about this study and asking him if he wishes to participate in your treatments. He will be asked to provide the study doctors at M. D. Anderson specific information about your treatments and any side effects you may have. All communications between your home doctor and your study doctors will be included as part of your M. D. Anderson medical record.

After the study ends, you will return for checkups every 3 months in the first year, every 4 months in Years 2 and 3, and every 6 months in Years 4 and 5. After that, checkups will be needed once a year. Blood (about 2 tablespoons) and bone marrow samples will be taken at these visits.

This is an investigational study. Ibritumomab tiuxetan and rituximab are approved by the FDA for commercial use. The other drugs used in the study are also approved for commercial use by the FDA. About 50 patients will take part in the study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high-risk Ann Arbor stage III-IV follicular lymphoma. High-risk is defined by advanced stage (III or IV), plus any 2 of the following features: age 60 or greater; elevated LDH; Hgb < 12; or number of involved nodal sites 5 or more .
2. Patients will be previously untreated.
3. Adequate organ function.
4. Follicular lymphoma, grade 3 (follicular large cell lymphoma): If eligible for a current large cell lymphoma protocol, that alternative protocol is recommended, particularly grade 3b or FLCL patients characterized as large non-cleaved cell. However, both FND and rituximab have established efficacy in FLCL, so if a patient is not eligible for a protocol for aggressive lymphoma (e.g., because of SCCL in the marrow), then registration on this trial is permitted.
5. Biopsy or fine-needle aspiration (FNA) material is strongly recommended for bcl-2 studies to verify rearrangement status of all patients who are designated "germline". (see section 6.4). For other patients, tissue availability is desirable but not mandatory.
6. Patients must have a performance status of Zubrod 3 or better
7. Patients must have adequate renal and hepatic function (creatinine < 2mg%; bilirubin < 2 mg%). Patients with renal or liver dysfunction due to organ infiltration by lymphoma may be eligible after discussion with the study chairman.
8. Patients may not receive other concurrent chemotherapy, radiotherapy, or immunotherapy.
9. Patients must sign an informed consent indicating that they are aware of the investigational nature of this study in keeping with the policies of the hospital.

Exclusion Criteria:

1. Patients who are unable or unlikely to be able to adhere to the treatment plan or to return to Houston for follow-up visits because of geographical, economic, emotional, or social considerations are not eligible for this study. Note: some follow-up care may be provided by outside physicians as long as the MD Anderson Cancer Center (MDACC) protocol for outside physician participation is strictly adhered to.
2. Patients with an absolute peripheral granulocyte count of < 1,000 and platelet count < 100,000 unless due to marrow infiltration or hypersplenism.
3. Patients with organ dysfunction, including bilirubin of > 2 mg% or serum creatinine level > 2 mg%, unless the alteration is due to lymphoma.
4. Patients with HIV infection should not be registered on this protocol.
5. Patients with an antecedent malignancy whose prognosis is poor (< 90% probability of surviving for 5 yrs).
6. All patients should have a cardiac ejection fraction of 50% or more by echocardiography or multiple gated acquisition scan (MUGA).
7. Patients who will not accept transfusions of blood products or supportive care measures such as antibiotics are not eligible for this study.
8. Female patients must not be pregnant or lactating, and men and women of reproductive potential must follow accepted birth control methods.
9. Patients who have received prior murine antibody therapy will be excluded.
10. Patients with evidence of active or prior infection of Hepatitis B are excluded. (Note: Persons vaccinated for Hepatitis B who have + antibodies are not excluded).

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2004-06-29 (Actual); Primary Completion 2021-02-12 (Actual); Study Completion 2021-02-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Fowler, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from June 2004 to May 2009.
Pre-assignment Details: Forty-nine patients with Follicular Lymphoma were enrolled in this single site, phase II trial. Two patients were removed after registration and did not start treatment: the first, due to physician's decision; the second, to pursue treatment at home.
Period: Overall Study
Arm/Group | R-FIND + Zevalin
Started | 49
No Treatment Per Protocol | 2
Toxicity Assessment | 47
Response Assessment | 45
Completed | 45
Not Completed | 4
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 62 [37 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 43
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 49
Bulky Disease [Count of Participants; unit: Participants]
  Bulky Disease >/=5 cm | 24
  No bulky disease | 25
Ann Arbor Stages [Count of Participants; unit: Participants] — I: involvement of a single lymph node region or of a single extralymphatic organ or site II: involvement of two or more lymph node regions on the same side of the diaphragm or localized involvement of an extralymphatic organ or site III: involvement of lymph node regions or structures on both sides of the diaphragmIV: diffuse or disseminated involvement of one or more extralymphatic organs, or either: isolated extralymphatic organ involvement without adjacent regional lymph node involvement, but with disease in distant sites involvement of the liver, bone marrow, pleura or cerebrospinal fluid
  Participants
    Ann Arbor Stage III | 7
    Ann Arbor Stage IV | 42
Follicular Lymphoma International Prognostic Index (FLIPI) [Count of Participants; unit: Participants] — A score indicating that a participant has 3 or more risk factors associated with follicular lymphoma and is considered in the high risk group.
  Participants
    FLIPI Score 3 | 40
    FLIPI Score 4 | 6
    FLIPI Score 5 | 2
Bone Marrow Biopsy [Count of Participants; unit: Participants]
  Bone Marrow Biopsy - Neg | 11
  Bone Marrow Biopsy - Pos | 37
Lactate Dehydrogenase (LDH) [Count of Participants; unit: Participants]
  LDH, units/ </= 618 | 35
  LDH, units/ >618 | 14
Beta 2 Microglobulin (B2M) [Count of Participants; unit: Participants]
  B2M, mg/l <2.2 | 15
  B2M, mg/l>/= 2.2 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Time to Progression (TTP)
Description: Regimen regarded as a success if median TTP can be prolonged to 36 months or greater. Time to Progression measured by the method of Kaplan and Meier, and accompanied by 95% confidence interval. Complete Response (CR) defined as those who achieve a normal state which includes no detectable evidence of disease on x-rays and Partial Response (PR) is defined as a 50% or more reduction in the sum of the products of the diameters of the 6 largest measurable lesions. No new sites of disease. av
Time Frame: baseline, 2 and 4 courses, approximately month 8, 9, and 12 months, then restaging every 4 months, then at 2 years every 4-6 months, then yearly until progressive disease or lost to follow up, average of 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 49
Participants
  Complete Response (CR) | 42
  Partial Response (PR) | 4

2. Secondary Outcome: Tolerance and Efficacy of Maintenance Therapy With Yttrium-90 Ibritumomab Tiuxetan (YIT)
Description: To assess the tolerance and efficacy of maintenance therapy with YIT. CR: defined as those who achieve a normal state which includes no detectable evidence of disease on x-rays. CRu: defined as "CR unconfirmed" on the basis of minimal residual abnormalities on x-ray such as a residual mass <25% of original measurement, and or residual indeterminate bone marrow aggregates. PR: a 50% or more reduction in the sum of the products of the diameters of the 6 largest measurable lesions. No new sites of disease. Progressive disease (PD) is also defined by the appearance of new lymph nodes, of other new or worsening sites of disease, such as > 50% increase in the size of liver and/or spleen, or a > 50% increase in absolute number of circulating lymphocytes.
Time Frame: cycle 1 and every 2 weeks thereafter until completion of therapy, an average of 10 years
Population: Participants that received YIT treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 38
Participants
  Complete Response (CR) | 37
  Progressive Disease | 1

3. Secondary Outcome: Tolerance and Efficacy of Maintenance Therapy With Rituximab
Description: To assess the tolerance and efficacy of maintenance therapy with rituximab. Participants proceeded to the rituximab maintenance program of 6 treatments comprising 1 every 2 months. CR: defined as those who achieve a normal state which includes no detectable evidence of disease on x-rays. CRu: defined as "CR unconfirmed" on the basis of minimal residual abnormalities on x-ray such as a residual mass <25% of original measurement, and or residual indeterminate bone marrow aggregates. PR: a 50% or more reduction in the sum of the products of the diameters of the 6 largest measurable lesions. No new sites of disease. Progressive disease (PD) is also defined by the appearance of new lymph nodes, of other new or worsening sites of disease, such as > 50% increase in the size of liver and/or spleen, or a > 50% increase in absolute number of circulating lymphocytes.
Time Frame: cycle 1 and every 2 weeks thereafter until completion of therapy, an average of 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 41
Participants
  Complete Response (CR) | 38
  Progression Disease (PD) | 3

4. Secondary Outcome: Median Progression Free Survival
Description: Progression-free survival time is defined as time from registration/randomization to the date of progression or death from any cause. Median Progression Free Survival estimated by the method of Kaplan and Meier, and accompanied by 95% confidence interval.
Time Frame: up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 47
months | 84 [67 to NA] — insufficient number of participants with events

5. Secondary Outcome: Progression Free Survival at 10 Years
Description: Progression-free survival time is defined as time from registration/randomization to the date of progression or death from any cause. PFS was estimated by the method of Kaplan and Meier, and accompanied by 95% confidence interval.
Time Frame: 10 years
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 47
months | 49 [37 to 66]

6. Secondary Outcome: Overall Survival
Description: OS is defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact. Median Overall Survival was estimated by the method of Kaplan and Meier, and accompanied by 95% confidence interval.
Time Frame: up to 5 years
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 47
months | 143 [143 to NA] — insufficient number of participants with events

7. Secondary Outcome: Percentage of Participants With Overall Survival Rate at 10 Years
Description: OS is defined as the interval from first dose of study treatment to the date of death, irrespective of the cause of death; subjects still alive will be censored at the date of the last contact. Overall Survival Rate estimated by the method of Kaplan and Meier.
Time Frame: 10 years
Measure: Number; unit: percentage of participants
Arm/Group | R-FIND + Zevalin
Number analyzed (Participants) | 47
percentage of participants | 69

ADVERSE EVENTS:
Time Frame: Adverse event reporting per patient done beginning at the start intervention per protocol through 30 days post intervention completion, up to 10 years
Arm/Group | R-FIND + Zevalin
All-Cause Mortality (participants affected / at risk) | 8/49
Serious Adverse Events (participants affected / at risk) | 34/49
Other Adverse Events (participants affected / at risk) | 46/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | R-FIND + Zevalin (N=49)
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 16
Anemia (Blood and lymphatic system disorders) | 1
Neutropenic Fever (General disorders) | 2
Secondary Malignancy (General disorders) | 2
Fatigue (General disorders) | 8
Pain (General disorders) | 6
Dyspnea (Cardiac disorders) | 5
Blurred Vision (Eye disorders) | 3
Dizziness (Nervous system disorders) | 3
Infection, normal ANC (Infections and infestations) | 3
Allergic reaction (Immune system disorders) | 2
Chest pain, non-cardiac (General disorders) | 2
Constipation (Gastrointestinal disorders) | 2
Edema, face (General disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Flushing (Immune system disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Rigors/chills (General disorders) | 1
Syncope (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | R-FIND + Zevalin (N=49)
Abdonimal distension (Gastrointestinal disorders) | 1
ALT increased (Metabolism and nutrition disorders) | 1
Allergic reaction (Immune system disorders) | 5
Allergic rhinitis (Immune system disorders) | 1
AST increased (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bilirubin increased (Investigations) | 1
Blurred Vision (Eye disorders) | 14
Bronchial infection (Infections and infestations) | 2
Bruising (Skin and subcutaneous tissue disorders) | 1
chills (General disorders) | 10
constipation (Gastrointestinal disorders) | 22
cough (Respiratory, thoracic and mediastinal disorders) | 6
creatinine increased (Investigations) | 2
diarrhea (Gastrointestinal disorders) | 18
dizziness (Nervous system disorders) | 18
dry skin (Skin and subcutaneous tissue disorders) | 1
dyspnea (Cardiac disorders) | 9
ear and labyrinth disorders - other (Eye disorders) | 1
Edema, face (General disorders) | 4
edema, limbs (General disorders) | 8
epistaxis (Blood and lymphatic system disorders) | 1
eye disorders- other (Eye disorders) | 11
fatigue (General disorders) | 18
fever (General disorders) | 11
flank pain (Musculoskeletal and connective tissue disorders) | 1
flatulence (Gastrointestinal disorders) | 1
flu like symptoms (General disorders) | 1
flushing (Skin and subcutaneous tissue disorders) | 1
gastritis (Gastrointestinal disorders) | 2
GI disorders- other (Gastrointestinal disorders) | 1
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
headache (Nervous system disorders) | 7
hiccups (Cardiac disorders) | 2
hyperglycemia (Metabolism and nutrition disorders) | 1
hyperuricemia (Metabolism and nutrition disorders) | 1
hypokalemia (Metabolism and nutrition disorders) | 1
hypotension (Cardiac disorders) | 2
infections other (Infections and infestations) | 7
insomnia (General disorders) | 3
irregular menstruation (Reproductive system and breast disorders) | 1
kyphosis (Musculoskeletal and connective tissue disorders) | 1
leukocytosis (Blood and lymphatic system disorders) | 3
lip infection (Infections and infestations) | 1
lung infection (Infections and infestations) | 1
lymphocyte count decrease (Blood and lymphatic system disorders) | 1
memory impairment (Nervous system disorders) | 10
mucosal infection (Infections and infestations) | 1
musositis oral (Gastrointestinal disorders) | 11
muculoskeletal and connective tissue disorder - other (Gastrointestinal disorders) | 1
myalgia (Musculoskeletal and connective tissue disorders) | 4
nausea (Gastrointestinal disorders) | 23
neoplasms (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
nervous systems disorders - other (Nervous system disorders) | 1
neutrophil count decreased (Blood and lymphatic system disorders) | 5
non-cardiac chest pain (General disorders) | 3
obstruction gastric (Gastrointestinal disorders) | 1
pain (General disorders) | 8
pain in extremity (General disorders) | 3
peripheral motor neuropathy (Musculoskeletal and connective tissue disorders) | 1
peripheral sensory neuropathy (Nervous system disorders) | 8
platelet count decreased (Blood and lymphatic system disorders) | 1
pruritus (Skin and subcutaneous tissue disorders) | 3
rash maculo-papular (Skin and subcutaneous tissue disorders) | 7
rectal pain (Gastrointestinal disorders) | 1
sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
skin disorders - other (Skin and subcutaneous tissue disorders) | 2
skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
skin infection (Skin and subcutaneous tissue disorders) | 1
somnolence (Nervous system disorders) | 1
sore throat (Respiratory, thoracic and mediastinal disorders) | 2
tremor (Nervous system disorders) | 1
urinary frequency (Renal and urinary disorders) | 1
urinary tract infection (Infections and infestations) | 1
urinary tract pain (Renal and urinary disorders) | 1
vomiting (Gastrointestinal disorders) | 6
watering eyes (Eye disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT00290511/Prot_SAP_000.pdf